CLINICAL TRIAL: NCT06439537
Title: Improving Consent In Trauma: Recall (ICIT: Recall) A Multicentre Study of Consent For Hip Fractures
Brief Title: ICIT: Recall A Multicentre Study of Consent For Hip Fractures
Acronym: ICIT: Recall
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC23137
Record Dates: First submitted 2024-05-06; First posted 2024-06-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Hip Fractures; Hip Injuries
Keywords: hip fracture; consent; incapacity
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single-group for all hip fracture patients: Single-group cohort for all hip fracture patients who are candidates for an operation
  Interventions: Other: Semi-structured questionnaire; Other: Post-operative interview

INTERVENTIONS:
Other: Semi-structured questionnaire — All patients recruited to the study will undergo a semi-structured questionnaire within 36 hours of admission
Other: Post-operative interview — All patients recruited to the study will undergo a semi-structured interview once they have reached post-operative day 7 or over

SUMMARY:
Hip fractures are a major cause litigation in patients undergoing trauma surgery. Common causes of litigation in hip operations are alleged incompetent surgery and development of pressure sources, both of which are associated with poor quality of consent. One aspect of poor consent is patients not being able to retain information discussed with them prior to their operation. There are many factors attributed to this, including pain in the acute setting, administration of sedating medications and the high rate of delirium in this patient cohort. However, even in individuals deemed to have capacity during the consent process, studies have shown that many were unable to explain what type of surgery they had or express knowledge of the potential complications. Importantly, the hip fracture patient demographic is very different from patients undergoing a planned procedure, in that they have had an acute injury following physical trauma, tend to be older and medically frailer. Research into the recall of patients undergoing gynaecological or abdominal surgeries further corroborate patients' poor recall of potential complications in the acute setting.

Patients with hip fractures face a range of risks, some of which can result in a substantial mortality rate regardless of whether surgery is performed. The list of complications includes infections in the hip joint and wound, development of pressure sores, occurrence of pulmonary embolism (PE) and deep vein thrombosis (DVT), myocardial infarction, urinary tract infection, pneumonia, and potential procedural failures. As such, the ability of patients to remember the discussed complications is critical to their well-being and overall quality of life and remains an unmet clinical need.

DETAILED DESCRIPTION:
Improving Consent In Trauma: Recall (ICIT Recall) will be a multicentre quality improvement project within the NHS clinical care setting. The aim of this study is to assess hip fracture patient's ability retain information regarding their injury, proposed operation, potential complications, and alternatives. following obtaining formal written consent. To that end, the project is intended to be a multicentre study, with interviews across a range of different health boards. The investigators also wish to listen to individual patients' experience of the surgical consent process through a follow-up interview once it has been over one week since their operation. Part (1), the structured face-to-face questionnaire was established to identify the extent of the problem and what patients find memorable or overlooked about the consent process. Part (2), the interview was designed to obtain qualitative data on what patients find important and to allow the participants to tell their story. The overarching objective of this project is to empower patients so that they are more involved and have a greater understanding of the operation that they have consented to. This includes simple measures such as providing a patient information leaflet or improving communication with the patient or close family members during their consent process. Sometimes, poor retention of information is unavoidable due to the significant pain and stress patients are under, and for this reason our aim is to improve the quality of consent for major procedures like hip operations.

As part of the project, the investigators also wish to engage with and capture patient-cantered experiences through a further interview. The investigators aim to like to capture their experience of the consent process entirely from the patient's perspective. Patient stories are a powerful tool to promote culture change in patient care. Unlike surveys, patient stories allow a seamless flow of thoughts and feelings that can provide insight into their journey to recovery. Here, the aim is to highlight the importance of good communication and an overall clear consent process in promoting wellbeing. This aspect of care tends to be overlooked. Addressing this issue is particularly important in delivering compassionate care within the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient on trauma and orthopaedic wards
* Is candidate for a hip fracture operation
* Able to provide informed consent
* Able to participate in a conversation (without the use of a translator)

Exclusion Criteria:

* Deemed to be too unwell or medically unstable to participate
* Under Adult With Incapacity Act or other detaining orders
* Patients scoring a 4AT score of 4 or more
* Unable to provide consent

Ages: 50 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants listed for hip fracture surgery, after sustaining a hip fracture surgery under the care of participating surgeons at the Royal Infirmary of Edinburgh. Approximately 100 participants will be included in this prospective cohort study recruited through consecutive sampling.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incapacity | Within 36 hours of admission
  Proportion of individuals admitted with hip fractures that do not have capacity to consent. The measurement tool will be the 4AT.
Retention of complications | Within 36 hours of admission
  Proportion of complications discussed initially in consenting individuals that were still retained by the time of interview (within 36 hours of admission).

SECONDARY OUTCOMES:
Thematic analysis of narrative contents | Post-operative day 7 to post-operative day 28
  The personal experience of giving consent for hip fracture operations through semi-structured questionnaires. The measurement tool is a thematic analysis using a qualitative coding framework, whereas the unit of measure is the frequency and prevalence of themes

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Clement, MBBS, MD, PhD, FRCS (T&O), Principal Investigator — NHS Lothian
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - NHS Lothian, Edinburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ring J, Talbot C, Cross C, Hinduja K. NHSLA litigation in hip fractures: Lessons learnt from NHSLA data. Injury. 2017 Aug;48(8):1853-1857. doi: 10.1016/j.injury.2017.06.009. Epub 2017 Jun 19. PMID 28648408
- [Background] Herrera-Perez M, Gonzalez-Martin D, Sanz EJ, Pais-Brito JL. Ethical Dilemmas with Regard to Elderly Patients with Hip Fracture: The Problem of Nonagenarians and Centenarians. J Clin Med. 2022 Mar 27;11(7):1851. doi: 10.3390/jcm11071851. PMID 35407459
- [Background] Zalmay P, Collis J, Wilson H. Patients Lacking the Capacity to Consent to Hip Fracture Surgery May Be Undergoing Major Operations Without Their Next of Kin Being Involved in Best-Interests Decisions: A Quality Improvement Report. Cureus. 2021 Dec 10;13(12):e20322. doi: 10.7759/cureus.20322. eCollection 2021 Dec. PMID 35028219
- [Background] Kalisvaart KJ, Vreeswijk R, de Jonghe JF, van der Ploeg T, van Gool WA, Eikelenboom P. Risk factors and prediction of postoperative delirium in elderly hip-surgery patients: implementation and validation of a medical risk factor model. J Am Geriatr Soc. 2006 May;54(5):817-22. doi: 10.1111/j.1532-5415.2006.00704.x. PMID 16696749
- [Background] Thiruchandran G, McKean AR, Rudran B, Imam MA, Yeong K, Hassan A. Improving consent in patients undergoing surgery for fractured neck of femur. Br J Hosp Med (Lond). 2018 May 2;79(5):284-287. doi: 10.12968/hmed.2018.79.5.284. PMID 29727232
- [Background] Probert N, Malik AA, Lovell ME. Surgery for fractured neck of femur - are patients adequately consented? Ann R Coll Surg Engl. 2007 Jan;89(1):66-9. doi: 10.1308/003588407X160846. PMID 17316526
- [Background] Bhangu A, Hood E, Datta A, Mangaleshkar S. Is informed consent effective in trauma patients? J Med Ethics. 2008 Nov;34(11):780-2. doi: 10.1136/jme.2008.024471. PMID 18974409
- [Background] Howard A, Webster J, Quinton N, Giannoudis PV. 'Hobson's choice': a qualitative study of consent in acute surgery. BMJ Open. 2020 Oct 8;10(10):e037657. doi: 10.1136/bmjopen-2020-037657. PMID 33033090